CLINICAL TRIAL: NCT01402063
Title: PPX and Concurrent Radiation for Newly Diagnosed Glioblastoma Without MGMT Methylation: A Randomized Phase II Study
Brief Title: PPX and Concurrent Radiation for Newly Diagnosed Glioblastoma Without MGMT Methylation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); Milton S. Hershey Medical Center (Other); University of Washington (Other); University of Massachusetts, Worcester (Other); MaineHealth (Other); University of California, San Diego (Other); Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, howard safran, Principal Investigator, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 244
Record Dates: First submitted 2011-07-08; First posted 2011-07-26 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Glioblastoma Multiforme
Keywords: Brain Tumors; Glioblastoma Multiforme; GBM
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — protein phosphatase 4; paclitaxel poliglumex; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radiation plus PPX(CT2103 (Experimental): Radiation therapy, Monday through Friday, for 6 weeks for a total of 30 treatments
  + intravenous PPX every week x 6 weeks for a total of 6 treatments
  Interventions: Drug: PPX (CT2103)
- radiation + Temozolomide (Active Comparator): Radiation therapy, Monday through Friday, for 6 weeks for a total of 30 treatments
  + Daily oral temozolomide(TMZ) (7 days) x 6 wks for a total of 42 days
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: PPX (CT2103) — XRT: 60 Gy at 2 Gy/fraction x 30 fractions PPX: 50 mg/m2/week x 6 weeks during radiation Temozolomide maintenance: Beginning 4 weeks after completion of chemoradiation, temozolomide d1-5 of 28 day cycle for 12 cycle maximum.
  Arms: radiation plus PPX(CT2103
Drug: Temozolomide — XRT: 60 Gy at 2 Gy/fraction x 30 fractions Temozolomide, 75 mg/m2/day, 7 days per week, from the first to the last day of radiotherapy Temozolomide maintenance: Beginning 4 weeks after completion of chemoradiation, temozolomide d1-5 of 28 day cycle for 12 cycle maximum
  Arms: radiation + Temozolomide

SUMMARY:
To obtain preliminary data in a randomized phase II study whether PPX/RT improves progression-free survival as compared to temozolomide/RT for patients with GBM without MGMT methylation.

DETAILED DESCRIPTION:
To evaluate the toxicities of PPX/RT To evaluate neuro-cognitive functional assessments of patients with GBM receiving PPX/RT To obtain preliminary data in a randomized phase II study whether PPX/RT improves overall survival as compared to temozolomide /RT for patients with GBM without MGMT methylation to facilitate planning a phase III study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of glioblastoma or gliosarcoma (WHO grade IV)
* GBM must have unmethylated MGMT as determined by central laboratory
* Diagnosis of GBM must be made by biopsy or surgical excision, either partial or complete; as long as there is sufficient tissue to determine MGMT status
* No prior chemotherapy or radiation for brain tumor
* Must be able to tolerate brain MRIs.

  *A diagnostic contrast-enhanced MRI must be performed postoperatively within 42 days prior to study registration.
* KPS >60.
* Age > 18
* Life expectancy of at least 3 months.
* Absolute neutrophil count > 1500/mm3, Platelets > 100,000/mm,
* Creatinine < 2 x ULN
* ALT or AST < 3 x upper limit of normal (ULN) and total bilirubin < 1.5x ULN.
* Patients with a prior history of low grade glioma who did not receive prior radiation or chemotherapy with transformation to grade IV brain tumor are eligible.
* Women must be non-lactating, and surgically sterile, post-menopausal or have a negative serum pregnancy test and agree to use adequate birth control. Males must agree to use adequate birth control.
* Voluntary, signed informed consent.

Exclusion Criteria:

* Acute infection or other medical condition that would impair study treatment
* No other active invasive malignancy unless disease free for at least 3 years.
* Prior temozolomide or PPX.
* Prior use of Gliadel wafers or any other intratumoral or intracavitary treatment are not permitted.
* Prior radiotherapy to the head or neck (except for T1 glottic cancer), resulting in overlap of radiation fields.
* No diffuse leptomeningeal disease, or gliomatosis cerebri.
* Use of any other experimental chemotherapy drug within the 60 days prior to randomization and during the trial. (Use of a non-chemotherapy investigational agent must be approved by the Brown University Oncology Group)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — BrUOG
Locations (9):
- United States (9):
  - UCSD Cancer Center, La Jolla, California
  - Maine Medical Center, Scarborough, Maine
  - UMASS Medical Center Cancer Center, Worcester, Massachusetts
  - SUNY Medical Center, Syracuse, New York
  - PSU, Hershey, Pennsylvania
  - Thomas Jefferson University Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - UT Southwestern Cancer Center, Dallas, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Jeyapalan S, Boxerman J, Donahue J, Goldman M, Kinsella T, Dipetrillo T, Evans D, Elinzano H, Constantinou M, Stopa E, Puthawala Y, Cielo D, Santaniello A, Oyelese A, Mantripragada K, Rosati K, Isdale D, Safran H; Brown University Oncology Group Study. Paclitaxel poliglumex, temozolomide, and radiation for newly diagnosed high-grade glioma: a Brown University Oncology Group Study. Am J Clin Oncol. 2014 Oct;37(5):444-9. doi: 10.1097/COC.0b013e31827de92b. PMID 23388562

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Plus PPX(CT2103: Radiation therapy, Monday through Friday, for 6 weeks for a total of 30 treatments
  + intravenous PPX every week x 6 weeks for a total of 6 treatments
  PPX (CT2103): XRT: 60 Gy at 2 Gy/fraction x 30 fractions PPX: 50 mg/m2/week x 6 weeks during radiation Temozolomide maintenance: Beginning 4 weeks after completion of chemoradiation, temozolomide d1-5 of 28 day cycle for 12 cycle maximum.
- Radiation + Temozolomide: Radiation therapy, Monday through Friday, for 6 weeks for a total of 30 treatments
  + Daily oral temozolomide(TMZ) (7 days) x 6 wks for a total of 42 days
  Temozolomide: XRT: 60 Gy at 2 Gy/fraction x 30 fractions Temozolomide, 75 mg/m2/day, 7 days per week, from the first to the last day of radiotherapy Temozolomide maintenance: Beginning 4 weeks after completion of chemoradiation, temozolomide d1-5 of 28 day cycle for 12 cycle maximum
Period: Overall Study
Arm/Group | Radiation Plus PPX(CT2103 | Radiation + Temozolomide
Started | 42 | 21
Completed | 39 | 18
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiation Plus PPX(CT2103 | Radiation + Temozolomide | Total
Number analyzed (Participants) | 42 | 21 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 15 | 42
  >=65 years | 15 | 6 | 21
Age, Continuous [Mean (Full Range); unit: years] | 62 [21 to 79] | 62 [49 to 82] | 62 [21 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 27 | 12 | 39
Region of Enrollment [Number; unit: participants]
  United States | 42 | 21 | 63

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival PPX/RT Versus TMZ/RT for Patients With GBM Without Methylation
Description: MRI response evaluated by RANO criteria
  * Complete Response (CR): Circumstance when the enhancing tumor is no longer seen by neuroimaging, with the patient off all steroids or on adrenal maintenance only; CR will be coded only if confirmed by a second CT/MR scan performed a minimum of 4 weeks after the initial scan coding a response.
  * Partial Response (PR): Decrease of > 50% in the product of two diameters. Patients should be receiving stable or decreasing doses of steroids. PR will be coded only if confirmed by a second CT/MR scan performed a minimum of 4 weeks after the initial scan.
  * Progression (P): A > 25% increase in tumor area (two diameters) provided that the patient has not had his/her dose of steroids decreased since the last evaluation period. This will not need a confirmatory scan. A concomitant decrease in steroid dose will rule out a progression designation during the first 2 months after completion of XRT.
Time Frame: Q 3 months on study then Q3 months in f/u for yr 1, q 4 months yr 2, q 6 months for approximately 4 ys.
Measure: Number; unit: participants
Arm/Group | Radiation Plus PPX(CT2103 | Radiation + Temozolomide
Number analyzed (Participants) | 42 | 21
participants | 31 | 15

ADVERSE EVENTS:
Time Frame: Baseline, throughout all treatment, at study discontinuation and 30 days post last dose of drug
Groups:
- Radiation Plus PPX and Maintenance: Radiation therapy, Monday through Friday, for 6 weeks for a total of 30 treatments
  + intravenous PPX every week x 6 weeks for a total of 6 treatments
  PPX (CT2103): XRT: 60 Gy at 2 Gy/fraction x 30 fractions PPX: 50 mg/m2/week x 6 weeks during radiation Temozolomide maintenance: Beginning 4 weeks after completion of chemoradiation, temozolomide d1-5 of 28 day cycle for 12 cycle maximum.
- Radiation + Temozolomide and Maintenance: Radiation therapy, Monday through Friday, for 6 weeks for a total of 30 treatments
  + Daily oral temozolomide(TMZ) (7 days) x 6 wks for a total of 42 days
  Temozolomide: XRT: 60 Gy at 2 Gy/fraction x 30 fractions Temozolomide, 75 mg/m2/day, 7 days per week, from the first to the last day of radiotherapy Temozolomide maintenance: Beginning 4 weeks after completion of chemoradiation, temozolomide d1-5 of 28 day cycle for 12 cycle maximum
Arm/Group | Radiation Plus PPX and Maintenance | Radiation + Temozolomide and Maintenance
Serious Adverse Events (participants affected / at risk) | 13/41 | 7/18
Other Adverse Events (participants affected / at risk) | 40/41 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Plus PPX and Maintenance (N=41) | Radiation + Temozolomide and Maintenance (N=18)
Anaphylactic Shock (Investigations) | 1 (1) | 0 (0)
Aspiration (Investigations) | 1 (1) | 0 (0)
Ataxia (Investigations) | 1 (1) | 0 (0)
Bowel Obstruction (Investigations) | 1 (1) | 0 (0)
Cardiac Event (Investigations) | 1 (1) | 0 (0)
Constipation (Investigations) | 1 (1) | 1 (1)
Dysphagia/Swallowing Difficulty (Investigations) | 1 (1) | 0 (0)
Dysphasia (Investigations) | 1 (1) | 0 (0)
Dyspnea/Shortness of Breath/COPD (Investigations) | 2 (2) | 0 (0)
Edema Cerebral/Brain Edema/Cerebral [Localized] Edema (Investigations) | 1 (1) | 0 (0)
Headache (Investigations) | 2 (2) | 1 (1)
Hemiparesis [Increasing] (LF Side) (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Investigations) | 2 (2) | 0 (0)
Hypocalcemia (Investigations) | 1 (1) | 0 (0)
Hypokalemia (Investigations) | 1 (1) | 0 (0)
Hypotension (Investigations) | 1 (1) | 0 (0)
Infection (Investigations) | 3 (5) | 0 (0) — (Infection normal ANC, COPD/bronchitis, Thrush (esophageal infection), pneumonia (URI), UTI, bacterial meningitis)
Loss of Balance (Investigations) | 1 (1) | 0 (0)
Lymphopenia/Lymphocytopenia/Decreased Lymphocyte Count/Lymphocyte # Decreased (Investigations) | 1 (2) | 0 (0)
Mental Status Changes (Investigations) | 6 (8) | 2 (2) — ( confusion/altered mental status, concentration impairment, cognitive decline, delirium)
Nausea/Increased Nausea/Nausea [Increasing] (Investigations) | 2 (2) | 2 (2)
Otitis (External)/ media/inflammation middle ear (Investigations) | 1 (1) | 0 (0)
Pain chest (Investigations) | 1 (1) | 0 (0)
Pulmonary Embolism (Investigations) | 1 (1) | 1 (1)
Seizure/Seizures (Investigations) | 2 (3) | 2 (3)
Stroke (Investigations) | 1 (1) | 0 (0)
Syncope (Investigations) | 1 (1) | 0 (0)
Thromboembolic Event (Investigations) | 1 (1) | 1 (1)
Vertigo (Investigations) | 1 (1) | 0 (0)
Vomitting (Investigations) | 1 (1) | 1 (1)
Weakness (generalized,proximal, LE proximal, LLE, Left UE and LE, arm) (Investigations) | 1 (1) | 0 (0)
PNEUMOPERITONEUM (Investigations) | 1 (1) | 0 (0)
WBC (Investigations) | 1 (1) | 0 (0)
SIADH (Investigations) | 1 (1) | 0 (0)
PLT (Investigations) | 1 (1) | 1 (1)
ANC (Investigations) | 1 (1) | 0 (0)
HCT (Investigations) | 1 (1) | 0 (0)
RBC (Investigations) | 1 (1) | 0 (0)
CSF elevated (Investigations) | 1 (1) | 0 (0)
Fever (Investigations) | 1 (2) | 0 (0)
Creatinine (Investigations) | 1 (1) | 0 (0)
Cough (Investigations) | 1 (1) | 0 (0)
Anemia (Investigations) | 1 (1) | 0 (0)
intratumoral hemorrhage (Investigations) | 0 (0) | 1 (1)
craniotomy (Investigations) | 0 (0) | 1 (1)
pancytopenia (Investigations) | 0 (0) | 1 (1)
pulseless electrical activity (Investigations) | 0 (0) | 1 (1)
Abdominal pain (Investigations) | 0 (0) | 1 (1)
Gallstones (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Plus PPX and Maintenance (N=41) | Radiation + Temozolomide and Maintenance (N=18)
abnormal blood prolactin (Investigations) | 1 (1) | 0 (0)
abrasions/lacerations: face, leg, finger (Investigations) | 3 (3) | 0 (0)
Acute gastroenteritis (Investigations) | 1 (1) | 0 (0)
Acne On Face and B/L Inguinal Region (Investigations) | 1 (1) | 0 (0)
Agitation (Investigations) | 2 (2) | 0 (0)
Akathisia (Investigations) | 3 (3) | 0 (0)
ALC Low/ALC Decreased (Investigations) | 3 (3) | 10 (10)
Alk Phos Elevated (Investigations) | 3 (3) | 0 (0)
Alopecia (Investigations) | 22 (22) | 3 (3)
Allergic reaction (Investigations) | 0 (0) | 1 (1)
LFTS (ALT/AST) (Investigations) | 6 (6) | 4 (4)
Ambulatory Dysfunction (Investigations) | 1 (1) | 0 (0)
Anemia (Investigations) | 13 (13) | 5 (5)
Anorexia/Decreased Appetite/Loss of Appetite (Investigations) | 11 (11) | 4 (4)
Anxiety/Anxiety [Increasing] (Investigations) | 6 (6) | 1 (2)
apathy (Investigations) | 0 (0) | 1 (1)
Aphasia (Investigations) | 4 (4) | 0 (0)
Aphasia (Motor) (Investigations) | 1 (1) | 0 (0)
Appetite (Increased) (Investigations) | 4 (4) | 0 (0)
Bells palsy (Investigations) | 0 (0) | 1 (1)
BILATERAL CAROTID BRUIT (Investigations) | 1 (1) | 0 (0)
Blurred Vision/Blurry Vision/homonymous hemianopsia(left)/cataracts/periorbital pressure (Investigations) | 16 (16) | 1 (1)
Bloody mucous (Investigations) | 0 (0) | 1 (1)
Bowel Incontinence (Investigations) | 1 (1) | 0 (0)
Bruising (Investigations) | 1 (1) | 0 (0)
BUN lab (Investigations) | 1 (1) | 0 (0)
CD4 Count Decreased (Investigations) | 3 (3) | 5 (5)
congestion/chest/ear (Investigations) | 4 (4) | 0 (0)
Chills (Investigations) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Investigations) | 1 (1) | 0 (0)
Cholesterol (Investigations) | 6 (6) | 0 (0)
Constipation (Investigations) | 9 (9) | 6 (6)
cough (Investigations) | 4 (4) | 1 (1)
cramping (Investigations) | 0 (0) | 1 (1)
creatinine (Investigations) | 4 (4) | 1 (1)
CSF elevated protein and collection (Investigations) | 1 (1) | 0 (0)
Cushingoid face (Investigations) | 4 (4) | 1 (1)
DARK LESION WITH IRREGULAR BORDERS - RIGHT MEDIAL ANKLE (BENIGN) (Investigations) | 1 (1) | 0 (0)
decreased arm swing (Investigations) | 6 (6) | 2 (2)
Dehydration (Investigations) | 5 (5) | 2 (2)
Depression (Investigations) | 5 (5) | 2 (2)
Dermatitis (Investigations) | 1 (1) | 2 (2)
Diarrhea (Investigations) | 5 (5) | 2 (2)
Dizziness (Investigations) | 10 (10) | 0 (0)
dry mouth (Investigations) | 2 (2) | 0 (0)
Dry skin (Investigations) | 1 (1) | 0 (0)
Dysphagia/Swallowing Difficulty (Investigations) | 2 (2) | 0 (0)
Dyspnea/Shortness of Breath (Investigations) | 7 (7) | 1 (1)
dysgeuisa (Investigations) | 2 (2) | 5 (5)
dyspepsia (Investigations) | 0 (0) | 1 (1)
Edema Cerebral/Brain Edema/Cerebral [Localized] Edema (Investigations) | 3 (3) | 0 (0)
Edema face/neck/hands (Investigations) | 1 (1) | 3 (3)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0)
erythema (Investigations) | 2 (2) | 1 (1)
Fatigue/Increased (Investigations) | 29 (29) | 16 (19) — Fatigue/Fatigue [Intermittent]/Fatigue [Increasing]/Fatigue (Worsening) - does not include somnolence
Facial Asymmetry (Investigations) | 2 (2) | 0 (0)
Fever (Investigations) | 4 (4) | 1 (1)
Flushing (Investigations) | 1 (1) | 0 (0)
flu like symptoms (Investigations) | 0 (0) | 1 (1)
Forehead trauma (Investigations) | 1 (1) | 0 (0)
fracture (Investigations) | 0 (0) | 1 (1)
Gait Unsteadiness/Unsteady Gait/proprioception/ cirumduction, motor deficit (Investigations) | 9 (9) | 1 (1)
GERD (Investigations) | 3 (3) | 0 (0)
Gum soarness (Investigations) | 1 (1) | 0 (0)
Hand Cramping (Investigations) | 3 (3) | 0 (0)
Hand tremor (Investigations) | 1 (1) | 0 (0)
Headache/Headache (Bifrontal)/Headache [Intermittent]/pressure (Investigations) | 17 (17) | 9 (9)
Hearing loss (Investigations) | 1 (1) | 0 (0)
Hernia (Investigations) | 0 (0) | 1 (1)
Hemorrhage (Intratumoral) (Investigations) | 1 (1) | 0 (0)
Hoarseness (Hoarse Voice) (Investigations) | 1 (1) | 0 (0)
Hypoalbuminemia (Investigations) | 1 (1) | 0 (0)
Hypocalcemia (Investigations) | 2 (2) | 1 (1)
Hyperglycemia (Investigations) | 14 (14) | 4 (4)
Hypoglycemia (Investigations) | 2 (2) | 0 (0)
hyperlipidemia (Investigations) | 0 (0) | 1 (1)
Hypertension (Investigations) | 1 (1) | 1 (1)
Hypotension (Investigations) | 1 (1) | 0 (0)
Hypertriglyceridemia (Investigations) | 2 (2) | 1 (1)
Hypokalemia (Investigations) | 10 (10) | 2 (2)
Hyperkalemia (Investigations) | 1 (1) | 0 (0)
Hypernatremia (Investigations) | 1 (1) | 0 (0)
Hypomagnesemia (Investigations) | 0 (0) | 1 (1)
Hypersensitivity to noise (Investigations) | 1 (1) | 0 (0)
Hyponatremia (Investigations) | 9 (9) | 2 (2)
Hypothyroidism (Investigations) | 1 (1) | 0 (0)
increased sputum (Investigations) | 1 (1) | 0 (0)
incisional tenderness (Investigations) | 0 (0) | 1 (1)
Infection (Investigations) | 15 (17) | 5 (5) — (Infection normal ANC, COPD/bronchitis, Thrush (esophageal infection), pneumonia (URI), UTI, bacterial meningitis, sinusitis)
Insomnia (Investigations) | 10 (10) | 5 (5)
Infusion Related Reaction (Investigations) | 1 (1) | 0 (0)
itchiness (Investigations) | 2 (2) | 0 (0)
intratumoral hemorrhage (Investigations) | 1 (1) | 0 (0)
jaw stiffness/tenderness (Investigations) | 0 (0) | 1 (1)
joint stiffness (Investigations) | 3 (3) | 0 (0)
Leukopenia (Investigations) | 10 (10) | 2 (2)
Lipase increase (Investigations) | 1 (1) | 0 (0)
Lower Extremity Edema (Bilateral)/ foot swelling (Investigations) | 6 (6) | 0 (0)
Lymphopenia/Lymphocytopenia/Decreased Lymphocyte Count/Lymphocyte # Decreased (Investigations) | 11 (11) | 6 (6)
Memory Loss (Worsening Short Term)/memory impairment (Investigations) | 7 (7) | 1 (1)
Mental Status Changes (Investigations) | 11 (11) | 1 (1) — ( confusion/altered mental status, concentration impairment, cognitive decline, delirium) (hallucination), (irritability)
mucous production increased (Investigations) | 0 (0) | 1 (1)
myopathy (Investigations) | 0 (0) | 1 (1)
narcolepsy (Investigations) | 1 (1) | 0 (0)
Nausea/Increased Nausea/Nausea [Increasing] (Investigations) | 21 (21) | 11 (11)
Neutropenia (Investigations) | 6 (6) | 3 (3)
Otitis (External)/ media/inflammation middle ear/tinnitus (Investigations) | 5 (5) | 0 (0)
Ear pain/pressure (Investigations) | 0 (0) | 1 (1)
Pain (Investigations) | 12 (17) | 5 (6) — (chest, leg, knee, hip/back,foot, LE, neck, body aches, general, incisional, shoulder, arm, lower back, abdomen, joint, schiatica)
Paresthesia (Hand)/LE/oral/neuropathy (Investigations) | 8 (8) | 2 (2)
PLTs (Investigations) | 17 (17) | 6 (6)
pain post herpatic neuralgia (Investigations) | 0 (0) | 1 (1)
Rash/skin irritation,seborrheic keratosis, desquamation of skin, maculopapular rash (Investigations) | 6 (6) | 4 (4)
pruritis (Investigations) | 0 (0) | 2 (2)
Psoriatic nails (Investigations) | 0 (0) | 1 (1)
Scrotal discomfort (Investigations) | 1 (1) | 0 (0)
Seizure/Seizures (Investigations) | 7 (7) | 1 (1)
sensory loss (Investigations) | 1 (1) | 0 (0)
sinusitis/post nasal (Investigations) | 0 (0) | 2 (2)
Skin lesions/ulceration (Investigations) | 2 (2) | 0 (0)
Somnolence (Investigations) | 1 (1) | 0 (0)
Swelling of Scalp [at Incision Site and Right Eyelid] (Investigations) | 1 (1) | 0 (0)
spasm extremity (Investigations) | 0 (0) | 1 (1)
Speech issues/vocal change (Investigations) | 2 (2) | 0 (0)
Stroke (Investigations) | 1 (1) | 0 (0)
Syncope (Investigations) | 1 (1) | 0 (0)
systolic murmur (Investigations) | 1 (1) | 0 (0)
Tachycardia (Sinus) (Investigations) | 3 (3) | 0 (0)
Tachypnea (Investigations) | 1 (1) | 0 (0)
Tooth ache (Investigations) | 1 (1) | 1 (1)
Tremor (Investigations) | 3 (3) | 0 (0)
Thromboembolic Event (Investigations) | 1 (1) | 0 (0)
ulcer (Investigations) | 0 (0) | 1 (1)
Urinary Incontinence (Investigations) | 2 (2) | 0 (0)
Urinary frequency (Investigations) | 3 (3) | 2 (2)
Wasting (General) (Investigations) | 1 (1) | 0 (0)
Watering eyes (Investigations) | 1 (1) | 1 (1)
Weakness (generalized,proximal, LE proximal, LLE, Left UE and LE, arm) (Investigations) | 15 (15) | 1 (1)
Weight Gain (Investigations) | 3 (3) | 1 (1)
Weight Loss (Investigations) | 5 (5) | 3 (3)
Wheezing (Investigations) | 1 (1) | 0 (0)
Vomiting (Investigations) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No